CLINICAL TRIAL: NCT06703996
Title: Bridging the Digital Divide of Wearables to Improve Health Outcomes and Quality of Life Among Black Prostate Cancer (CaP) Survivors
Brief Title: InBody Band 3 Fitness Tracker to Improve Health Outcomes and Quality of Life in Black Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emma Fortune Ngufor, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-009203; NCI-2024-09282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-009203 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-11-15; First posted 2024-11-25 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (InBody Band 3 fitness tracker) (Experimental): Patients wear the InBody Band 3 fitness tracker continuously and participate in check-in/goal-setting discussions over 20-30 minutes weekly for 6 weeks.
  Interventions: Other: Discussion; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Discussion — Participate in check-in/goal-setting discussions
  Other Names: Discuss
Other: Medical Device Usage and Evaluation — Wear the InBody Band 3 fitness tracker
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well the InBody Band 3 fitness tracker works to improve physical activity, body composition, and quality of life in Black prostate cancer survivors. Prostate cancer is the most common cancer in men and Black men are more likely to be diagnosed with prostate cancer in an advanced stage. Body composition is associated with disease progression, treatment response, and survival in cancer patients. Reducing stress and maintaining healthy levels of physical activity and sleep are important for a healthy body and improving outcomes, however, there is currently little evidence available on the physical activity, stress levels and sleep patterns in this population. Wearable health activity trackers and smart watches are tools that can be used to track physical activity, stress, sleep and body composition and have been shown to have a positive impact in many patient populations. The InBody Band 3 may be an effective method to improve physical activity, body composition and quality of life in Black prostate cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of a remote wearables-based intervention among Black prostate cancer survivors.

II. Assess the acceptability of the wearables-based intervention among Black prostate cancer survivors.

OUTLINE:

Patients wear the InBody Band 3 fitness tracker continuously and participate in check-in/goal-setting discussions over 20-30 minutes weekly for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to read/speak English and are able to communicate by phone
* 18 years of age or older
* Self-identify as Black
* Have been diagnosed with stage I-IV prostate cancer
* Have an active email address and are able to regularly check emails for electronic surveys
* Own and are willing to use a personal smartphone with regular/reliable access to the internet to sync regularly with a fitness tracker
* Are willing to wear and use a smart fitness tracker for 6 weeks and allow sharing of their fitness data with the study team
* Are not currently undergoing adjunct cancer therapy (e.g. chemotherapy, radiation) during the 6 weeks of study participation, except oral tyrosine kinase inhibitor or hormonal therapies; and
* Are an existing Mayo patient
* Self-report that they would like to improve their physical activity during initial study coordinator contact

Exclusion Criteria:

* Live outside of the United States (U.S)
* Have an implanted medical device (e.g., pacemaker, etc.) or a life-sustaining device (e.g., patient monitoring device)
* Have a self-reported history of a psychiatric disorder(s) or moderate to severe cognitive impairment precluding participation in the study intervention or preventing the ability to provide independent informed consent
* Are on prolonged bed rest (i.e., more than half of the waking day in bed) by self-report
* Currently have any lower extremity injury that impedes them from engaging in walking for one block
* Are unable to walk for at least one block without a walking aide by self-report; or
* Regularly use a wheelchair for mobility by self-report

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Adherence rate | Up to 6 weeks
  The adherence rate will be calculated as the ratio of number of valid data collection weeks to the number of expected valid data collection weeks for each participant. A group average adherence rate of 80% will be considered feasible.
Change in acceptability scale score | Up to 8 weeks
  Will be assessed using the 6-item Acceptability survey for physical activity interventions. Participants will be asked to rate each question from 0 (not at all) to 10 (extremely), and a mean score will be calculated. An average group rating of 8.0 or higher on a 10-point scale will be required to determine intervention acceptability. Change in score will be defined as the final intervention week's value minus the first week's value.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Fortune Ngufor, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials